CLINICAL TRIAL: NCT05667844
Title: Effects of Mind-body Exercises in a Patient With Mood Disorders: a Case Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Karoline Almeida Pereira, Master of science student, Universidade Federal do Rio de Janeiro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IPUBCDA
Record Dates: First submitted 2022-11-29; First posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Mood Disorders; Mind-body Exercise
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Intervention Model Description: Study case
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mind-body intervention (Experimental)
  Interventions: Behavioral: interoceptive mind-body exercise

INTERVENTIONS:
Behavioral: interoceptive mind-body exercise — A interoceptive mind-body exercise program in a patient with Generalized Anxiety Disorder and Major Depressive Disorder based on a Multidimensional Assessment of Interoceptive Awareness. Each session of the body-mind intervention lasts 80 minutes and is supervised by physical education professionals. The intervention is divided in 4 parts, that are: Preparatory phase (reception) the subjects will be welcomed through subjective analyzes of the researcher; Initial phase (preliminares) Mindfulness, grounding, sensory stimulation and joint warm-up exercises are performed; main phase (exercises) stretching, mobility, posture and balance exercises are performed with full attention and listening after each exercise; Final phase (relaxation) breathing exercises, stretching exercises, body scanning and relaxation are performed.

SUMMARY:
The interoception capacity may be changed with mind-body intervention. This study case investigated the interoceptive capacity, measured by MAIA scale of a pacient with mood disorders and if it can be influenced through of a 7 weeks intervention of interoceptive exercises and the impaction in the patient´s daily life. The aim was analyse the effects of mind-body exercise program with interoceptive approach in the anxiety and depression symptoms, interoceptive capacity, as well your impact in paitient's daily activities. M.S is 47 years old, was forwarded from University Hospital Clementino Fraga Filho to extension project named as "corpo&mente" (body-mind), an anamnesis was performed including patient's life story, interoceptive scale, anxiety and depression scale from Hamilton and a risk stratification to realize physical activities (it was also performed post-intervention). The exercise program lasted 1h 15 min and it was performed once a week.

ELIGIBILITY:
Inclusion Criteria:

* Participants with anxiety or/and depression clinical diagnosis
* Participants who do not do formal meditation practices

Exclusion Criteria:

* Participants with other diagnosis
* Patients with cognitive conditions

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Mnteroceptive capacity | Day 1
  assessed by interoceptive scale named Multidimensional Assessment of Interoceptive Awareness. In this scale, the average of each of the seven dimensions is calculated, the higher the value, the greater the interoceptive capacity.
Anxiety symptoms | Day 1 and after 7 weeks
  To measure the level of anxiety symptoms the Hamilton Anxiety scale was performed. The Hamilton Anxiety Scale has 14 items, each item is scored from 0 (absent symptoms) to 4 (disabling symptoms(, The higher the scores, the greater the levels of anxiety.
Depression symptons | Day 1 and after 7 weeks
  Hamilton Depression was used to measure the level of depression symptons. It has 21 items, where the scores for symptoms from 0 to 5. The higher the scores, the greater the levels of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No